CLINICAL TRIAL: NCT03141762
Title: Understanding the Impact of Critical Illness on Falls Risk - a 12 Month Observational Study
Status: Completed | Type: Observational
Sponsor: University of Melbourne (Other)
Collaborators: Melbourne Health (Other); University of Kentucky (Other)
Responsible Party: Principal Investigator, Selina M Parry, Chief Investigator, University of Melbourne
Other Study IDs: 2016.365
Record Dates: First submitted 2017-04-10; First posted 2017-05-05 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Critical Illness
Keywords: Falls; Intensive care
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Understanding the Impact of Critical Illness on Falls Risk - a 12 Month Observational Study

DETAILED DESCRIPTION:
This observational study aims to investigate the incidence and risk factors for falls in the first 12 months post hospital discharge in patients following an ICU admission. It also aims to determine factors at hospital discharge which may predict future falls risk at 12 months and examine the physical activity levels of ICU survivors. Furthermore, it also will investigate the relationship between falls, fear of falling and activity limitations and participation restriction. All adult patients in intensive care that have been mechanically ventilated for over 48 hours, and remain in the ICU at least 4 days will be considered for inclusion. The primary outcome measure is a 12 month falls diary which commences on hospital discharge. There will also be Physiotherapy assessments just prior to hospital discharge, 3, 6, and 12 months post hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* hospitalised adults aged 18 years
* with an ICU admission requiring invasive mechanical ventilation for at least 48 hours and remain in ICU > 4 days

Exclusion Criteria:

* Pregnant
* Insufficient English language skills to read and understand questionnaires and patient information consent form
* Pre-existing documented cognitive impairment
* Spinal cord injury or other primary neuromuscular disease or new brain injury
* Patient unable to be followed up due to geographic location
* New lower limb fracture on this admission
* Liver failure with abdominal distension due to ascites requiring fortnightly drainage
* Recent history of stroke or major surgery affecting lower limb e.g. Total knee or hip replacement in the past 12 weeks
* Neurological disorders such as Parkinson disease or multiple sclerosis
* Poor premorbid function defined as <10 metres ambulation +/- gait aid independently
* Frequent falls history defined as 3 or more falls over 2 months
* incarcerated or safety concerns for follow up
* discharged to palliative hospice facility
* not expected to survive to 3 months post hospital discharge
* unable to provide informed consent before hospital discharge due to current cognitive state (e.g. delirium, psychosis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will include: hospitalised adults aged 18 years and above with an ICU admission requiring invasive mechanical ventilation for at least 48 hours.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-05-03 (Actual); Primary Completion 2020-09-20 (Actual); Study Completion 2020-09-20 (Actual)

PRIMARY OUTCOMES:
Falls calendar - number of falls per month for 12 months, self-recorded by participant | One per month for 12 months
  12-monthly falls calendar - This will record time to first fall, falls, incidence, number of falls including injurious falls.

SECONDARY OUTCOMES:
Muscle ultrasound imaging | Baseline, 3, 6, and 12 months post discharge
  Ultrasound of rectus femoris and tibialis anterior
Hand held dynamometry | Baseline, 3, 6, and 12 months post discharge
  Muscle strength
mini-BEST | Baseline, 3, 6, and 12 months post discharge
  Balance
4 metre walk test | Baseline, 3, 6, and 12 months post discharge
  Gait
MoCA | Baseline, 3, 6, and 12 months post discharge
  Cognitive
Physical activity levels | Baseline, 3, 6, and 12 months post discharge
  Physical activity as measured as per title. Assessed using a physical activity tracker that participants will wear.
Clinical frailty scale questionairre | Baseline, 3, 6, and 12 months post discharge
  Frailty
Falls Risk for Older People in the Community Setting (FROP-com) Questionairre | 3, 6, and 12 months post discharge
  Falls risk
Fall efficacy scale questionnaire (version: FES-International short form) | Baseline, 3, 6, and 12 months post discharge
  Individuals are asked to rate, on a four-point Likert scale, their concerns about the possibility of falling when performing 16 activities.
Hospital Anxiety and Depression Scale (HADS) Questionairre | Baseline, 3, 6, and 12 months post discharge
  It is a self-rating scale that measures anxiety and depression in both hospital and community settings.
EuroQol five dimensions questionnaire (version: EQ-5D-5L) | Baseline, 3, 6, and 12 months post discharge
  Self-reported health-related quality of life questionnaire.
Impact of Event Scale questionnaire (version: IES-R) | Baseline, 3, 6, and 12 months post discharge
  It is a self-reported questionnaire that measures It measures the severity of intrusion, avoidance, and hypervigilance symptoms, experienced over the past week.
Short Physical Performance Battery | Baseline, 3, 6, and 12 months post discharge
  physical test evaluation of balance, strength, and walking ability
Healthcare usage | 3, 6, and 12 months post discharge
  Categorise readmissions and what health services are used post hospital discharge
FACIT Fatigue Scale (in subgroup) | 3, 6 and 12 months
  Fatigue levels self report questionnaire
Sedentary behaviour questionnaire (in subgroup) | 3, 6, and 12 months
  Weekend and weekday questionnaire of sedentary behaviour in hours
Conor Davidson Resilience Questionnaire (in subgroup) | 3, 6, and 12 months
  self report resilience questionnaire
Life Orientation Revised Optimism Scale (in subgroup) | 3, 6, and 12 months
  10 item self report optimism scale, higher scores indicate higher optimism
Pittsburgh Sleep Quality Index (in subgroup) | 3, 6, and 12 months
  questionnaire that evaluates sleep quality, higher scores indicate poorer sleep
MYMOP2 (in subgroup) | 3, 6, and 12 months
  short questionnaire which asks patients to rate their top problems and activity limitations
Memorial symptoms questionnaire short form | 3, 6, and 12 months
  questionnaire which covers different symptoms and how much it bothers the patient on a likert scale
Return to work | 3, 6 and 12 months
  questionnaire which provides time to return to work and impact on finances

CONTACTS AND LOCATIONS:
Overall Officials: Selina Parry, PhD, Principal Investigator — University of Melbourne
Locations (2):
- UK Healthcare, Lexington, Kentucky, United States
- Melbourne Health, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
Currently undecided if plan to make IPD available will update the Clinical Trials Registry.